CLINICAL TRIAL: NCT07029568
Title: A First in Human Dose Study to Assess the Safety, Tolerability, Pharmacokinetics, and Target Engagement of Single and Multiple Oral Administrations of NNC0705-0001 in Healthy Adults
Brief Title: A Study to See How Safe a New Medicine (NNC0705-0001) is in Healthy People
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NN6705-8141; U1111-1315-6842 (Other: World Health Organization); 2024-519478-38 (Other: European Medical Agency (EMA))
Record Dates: First submitted 2025-06-11; First posted 2025-06-19 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Healthy Volunteers; Chronic Kidney Disease
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Sponsor staff involved in the clinical trial is masked according to company standard procedures.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Part A: NNC0705-0001 (Experimental): Participants will receive 6 different single ascending doses of NNC0705-0001 via oral administration.
  Interventions: Drug: NNC0705-0001
- Part A: Placebo (Placebo Comparator): Participants will receive single ascending dose of placebo matching NNC0705-0001 via oral administration.
  Interventions: Drug: Placebo
- Part B: NNC0705-0001 (Experimental): Participants will receive 4 different multiple ascending doses of NNC0705-0001 via oral administration.
  Interventions: Drug: NNC0705-0001
- Part B: Placebo (Placebo Comparator): Participants will receive multiple ascending doses of placebo matching NNC0705-0001 via oral administration.
  Interventions: Drug: Placebo
- Part C: NNC0705-0001 (Experimental): Participants will receive 2 separate single doses of NNC0705-0001 at a previously safety-cleared dose level in PART A, either in a fed or fasted state.
  Interventions: Drug: NNC0705-0001

INTERVENTIONS:
Drug: NNC0705-0001 — NNC0705-0001 will be administered orally.
  Arms: Part A: NNC0705-0001; Part B: NNC0705-0001; Part C: NNC0705-0001
Drug: Placebo — Placebo matching NNC0705-0001 will be administered orally.
  Arms: Part A: Placebo; Part B: Placebo

SUMMARY:
The study is testing a new study medicine (called NNC0705-0001), as a potential medicine to treat chronic systemic inflammation, which is known for increasing the risk of developing cardiometabolic diseases. The aim of this study is to see if the study medicine is safe, how it works in our body, and what our body does to the study medicine. The participant will either get NNC0705-0001 or placebo (a "dummy medicine" without the active ingredient). Which treatment the participant gets is decided by chance. The study consists of 3 parts: PART A - single ascending dose (SAD); PART B - multiple ascending doses (MAD) and PART C - food effect (FE) on the pharmacokinetic (PK) properties of NNC0705-0001 and will last about 35 days (PART A) and 41 days (PART B and C).

ELIGIBILITY:
Inclusion Criteria:

* Men, or women of non-childbearing potential.
* Age 18-55 years (both inclusive) at the time of signing the informed consent.
* Body mass index (BMI) between 18.5 to 29.9 kilogram per meter square (kg/m^2) (both inclusive) at screening.
* Body weight: greater than or equal to (≥) 50 kilogram (kg) at screening.
* Considered to be generally healthy based on the medical history, physical examination, and the results of vital signs, electrocardiogram and clinical laboratory tests performed during the screening visit, as judged by the investigator.

Exclusion Criteria:

* Known or suspected hypersensitivity to study intervention(s) or related products.
* Any condition, which in the investigator's opinion might jeopardise participant's safety or compliance with the protocol.
* Any of the below laboratory safety parameters at screening outside normal range, see designated reference range documents for specific values; Alanine Aminotransferase (ALT) greater than (>) Upper limit of normal (ULN); Aspartate aminotransferase (AST) > ULN; Total Bilirubin (BIL) > ULN; Creatinine > ULN; International normalized ratio (INR) > ULN; High-Sensitivity C-Reactive Protein (hsCRP) > 5 milligram per liter (mg/L) (males) and > 8 mg/L (females)
* Use of prescription medicinal products or vaccines within 14 days before dosing and/or non-prescription medicinal products within 7 days before dosing. Exceptions are: Topical medications not reaching systemic circulation; less than once per week of over the counter paracetamol and/or acetylsalicylic acid at their labelled doses for mild pain; vitamins at their labelled doses.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 116 (Actual)
Dates: Start 2025-06-13 (Actual); Primary Completion 2025-12-10 (Actual); Study Completion 2025-12-10 (Actual)

PRIMARY OUTCOMES:
PART A: Number of treatment emergent adverse events (TEAE) | From time of dosing (day 1) to end of study (day 7)
  Measured in number of events.
PART B: Number of TEAEs | From time of dosing (day 1) to end of study (day 13)
  Measured in number of events.
AUC, SD; the area under the NNC0705-0001 plasma concentration-time curve after a single dose | From pre-dose (day 1 or day 8) to day 2 or day 9
  Measured in Hour x Micromole (hr×μM).

SECONDARY OUTCOMES:
PART A: AUC0-t, SD; the area under the NN0705-0001 plasma concentration-time curve from time 0 to last measurable plasma concentration after a single dose | From pre-dose (day 1) to day 5
  Measured in hr×μM.
PART A: AUC0-∞, SD; the area under the NNC0705-0001 plasma concentration-time curve from time 0 to infinity after a single dose | From pre-dose (day 1) to day 5
  Measured in hr×μM.
PART A: Cmax, SD; the maximum plasma concentration of NNC0705-0001 after a single dose | From pre-dose (day 1) to day 5
  Measured in micromole (μM).
PART B: AUCtau, MD; the area under the NN0705-0001 plasma concentration-time curve from time 0 to tau after the last dose | From pre-dose (day 7) to end of study (day 13)
  Measured in hr×μM.
PART B: Cmax, MD; the maximum plasma concentration of NNC0705-0001 after last dose | From pre-dose (day 7) to end of study (day 13)
  Measured in μM.
PART C: Cmax, SD; the maximum plasma concentration of NNC0705-0001 after a single dose | From pre-dose (day 1 or day 8) to day 2 or day 9
  Measured in μM.
PART C: Number of TEAEs | From time of dosing (day 1) to end of study (day 12)
  Measured in number of events.

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Transparency (dept. 2834), Study Director — Novo Nordisk A/S
Locations (1):
- ICON - location Groningen, Groningen, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk disclosure commitment on novonordisk-trials.com
URL: https://novonordisk-trials.com